CLINICAL TRIAL: NCT07407556
Title: Exploring the Use of Genetic and Behavioural Data in Tailoring Dietary and Lifestyle Support: An n=1 Randomised Trial
Brief Title: Exploring the Use of Genetic and Behavioural Data in Tailoring Dietary and Lifestyle Support
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandra King (Other)
Collaborators: Optimyse Nutrition LTD (Unknown)
Responsible Party: Sponsor-Investigator, Alexandra King, Head of School Allied Health and Life Sciences, St. Mary's University, Twickenham
Organization: St. Mary's University, Twickenham (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SMU_ETHICS_2025-26_195
Record Dates: First submitted 2026-01-23; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Adherence to a Personalised Nutrition Programme
Keywords: personalised nutrition; behaviour change; adherence

STUDY DESIGN:
Intervention Model Description: This study is a 6-week n-of-1 micro-randomised trial (MRT) across multiple participants designed to evaluate the effect of message tailoring (psychology-tailored vs neutral) on short-term habit adherence within a fully personalised lifestyle intervention. An MRT is a within-person experimental design in which each participant is repeatedly randomised to different intervention conditions. This allows estimation of causal, moment-level effects even in small samples because each participant serves as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static personalisation (Active Comparator): All participants receive a fully personalised dietary and lifestyle plan based on:
  * baseline lifestyle and diet
  * health status
  * environmental context
  * genetic polymorphisms (e.g., FTO, APOA2, TCF7L2, CLOCK, TMPRSS6, FADS1/2, MTNR1B, CYP1A2, taste receptors) This ensures that both study arms receive personalised nutrition, reflecting current best practice.
  Participants receive:
  * One fixed daily behaviour goal, aligned with the weekly pillar
  * Personalised only according to diet, lifestyle, health status and genetics
  * Delivered at a pre-selected time chosen by the participant (e.g., 8:30-10:00)
  No adaptation is made based on:
  * psychological traits
  * daily mood/energy
  * anticipated or reported barriers
  * communication preferences (tone, length, mode) This reflects current "gold standard" personalised nutrition: personalised by biology and lifestyle, but not by psychology or dynamic states.
  Interventions: Behavioral: Neutral message
- Fully personalised (Experimental): All participants receive a fully personalised dietary and lifestyle plan based on:
  * baseline lifestyle and diet
  * health status
  * environmental context
  * genetic polymorphisms (e.g., FTO, APOA2, TCF7L2, CLOCK, TMPRSS6, FADS1/2, MTNR1B, CYP1A2, taste receptors) This ensures that both study arms receive personalised nutrition, reflecting current best practice.
  Participants receive the same nutritional and lifestyle content, but daily goals are adapted based on:
  Stable Traits
  * Big Five personality
  * Health locus of control
  * Optimism bias
  * Delay discounting
  * Self-determination
  * Stress/anxiety baseline
  * Habit awareness
  * Values/motivations
  * Reward preferences Daily State
  * Morning energy rating (1-5)
  * Expected barriers
  * Context (home vs office vs weekend) Communication Preferences
  * tone (coachy, compassionate, factual, brief)
  * message length (low/medium/high)
  * mode (text, voice, image) Environmental and Social Context (e.g., Friday office snacks, partner-driven late dinners)
  Interventions: Behavioral: Psychology-tailored message

INTERVENTIONS:
Behavioral: Psychology-tailored message — Participants receive the same nutritional and lifestyle content, but daily goals are adapted based on:
  Stable Traits
  * Big Five personality
  * Health locus of control
  * Optimism bias
  * Delay discounting
  * Self-determination
  * Stress/anxiety baseline
  * Habit awareness
  * Values/motivations
  * Reward preferences Daily State
  * Morning energy rating (1-5)
  * Expected barriers
  * Context (home vs office vs weekend) Communication Preferences
  * tone (coachy, compassionate, factual, brief)
  * message length (low/medium/high)
  * mode (text, voice, image) Environmental and Social Context (e.g., Friday office snacks, partner-driven late dinners)
  Daily personalisation influences:
  * difficulty level of the daily goal
  * specific behaviour change technique (BCT) chosen (e.g., action planning vs implementation intention vs coping planning)
  * tone, structure and timing of the message
  * reinforcement style The nutrition content remains identical; only HOW it is delivered changes.
  Arms: Fully personalised
Behavioral: Neutral message — Participants receive:
  * One fixed daily behaviour goal, aligned with the weekly pillar
  * Personalised only according to diet, lifestyle, health status and genetics
  * Delivered at a pre-selected time chosen by the participant (e.g., 8:30-10:00)
  No adaptation is made based on:
  * psychological traits
  * daily mood/energy
  * anticipated or reported barriers
  * communication preferences (tone, length, mode) This reflects current "gold standard" personalised nutrition: personalised by biology and lifestyle, but not by psychology or dynamic states.
  Arms: Static personalisation

SUMMARY:
Personalised nutrition approaches typically rely on static information such as health status, lifestyle and genetic data. However, adherence often remains low because daily behaviours are influenced by psychological states, motivation and real-time barriers. There is growing interest in whether integrating behavioural signals and timely prompts could strengthen engagement. The purpose of this study is to explore whether incorporating psychological adaptation and just-in-time behavioural prompts leads to better adherence to a personalised nutrition programme compared with commonly used personalised approach (combining health, lifestyle and genetics data without psycho-behavioural adaptation). Using a six-week n-of-1 randomised trial design implemented across multiple participants, the research will also assess the feasibility of delivering this adaptive support in a free-living environment, as well as participants' engagement, acceptability and perceived usefulness. These findings will inform the development of an adaptive personalised nutrition AI agent.

ELIGIBILITY:
Inclusion Criteria:

* Participants must:

  1. Be 18-45 years old.
  2. Have a BMI between 18.5 and 40 kg/m² (normal weight to obesity categories).
  3. Own a smartphone with WhatsApp installed.
  4. Be willing to receive daily messages for 6 weeks.
  5. Be able to provide informed consent.
  6. Be willing to provide a cheek swab for DNA analysis.
  7. Have sufficient English proficiency to understand daily written instructions.

Given that the programme focuses on the six pillars of lifestyle medicine (nutrition, physical activity, sleep, stress management, social connection, and alcohol/substance moderation), participants must be able to safely engage with light lifestyle recommendations.

Exclusion Criteria:

* Participants will be excluded if they:

  1. Have a diagnosed eating disorder or significant disordered eating symptoms.
  2. Are currently pregnant or breastfeeding.
  3. Have any medical condition requiring medically supervised dietary modification (e.g., diabetes requiring medication, kidney disease, coeliac disease).
  4. Are currently taking medication that significantly affects appetite, weight, or metabolism (e.g., GLP-1 agonists).
  5. Work night shifts
  6. Have severe mental health conditions (e.g., moderate-severe depression, psychosis).
  7. Are participating in another behaviour-change or weight-related study.
  8. Are unwilling to receive WhatsApp messages
  9. Are unwilling to receive genetic information This will be checked with PARQ questionnaire

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Adherence | From enrolment to the end of the 6 week intervention
  Adherence is defined as daily completion or active attempt of the assigned lifestyle goal. Adherence is measured using a brief daily self-report item delivered via WhatsApp as part of an ecological momentary assessment. Each day, participants are asked whether they completed or actively attempted the assigned goal (Yes/No). Daily adherence is coded as a binary outcome (1 = completed, 0 = not completed). Adherence rates are calculated as the proportion of completed goal days relative to total analysable person-days and compared between personalised intervention days and static control days. An analysable person-day is defined as a day on which a goal message was successfully delivered and a corresponding adherence response was received within the response window. Days with missing responses or delivery failures are excluded from adherence analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's University, Twickenham, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The findings will be used to develop a commercial App for dietary behaviour change